CLINICAL TRIAL: NCT04589390
Title: Selexipag for the Treatment of Schistosomiasis-Associated Pulmonary Arterial Hypertension
Acronym: SELSCH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAP129
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Hypertension; Schistosomiasis
Keywords: pulmonary arterial hypertension; schistosomiasis; selexipag; treatment; efficacy; safety
MeSH Terms: conditions — Hypertension, Pulmonary; Schistosomiasis; Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Intervention Model Description: Evaluation of hemodynamics and surrogate markers (clinical variables, BNP levels, six-minute walking test distance, and heat shock protein 70 levels) before and after the introduction of selexipag for the treatment of schistosomiasis-associated pulmonary arterial hypertension patients, that were already receiving at least one therapy for pulmonary arterial hypertension, excluding other drugs from the prostacyclin pathway.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selexipag (Other): Selexipag will be up titrated for a period that will last 12 weeks (Phase 2). The initial dose will be 200 mcg of selexipag every 12 hours, with weekly dose increases of 200 mcg, up to the maximum dose of 1600 mcg every 12 hours or until the classic side effects of the prostacyclin pathway drugs (headache, mandibular pain), among others) arise. The dose will then be reduced by 200 mcg per dose, and this will be the maximum dose considered for that particular patient, maintained in Phase 3 (16 weeks).
  Interventions: Drug: Selexipag

INTERVENTIONS:
Drug: Selexipag — treatment with selexipag

SUMMARY:
Pulmonary arterial hypertension (PAH) is a severe, progressive and potentially fatal disease that impairs the pulmonary circulation and leads to right ventricular failure. One of the world most prevalent etiologies of PAH is schistosomiasis-associated pulmonary arterial hypertension (Sch-PAH). New drugs have emerged to treat other forms of PAH, but their benefits cannot be automatically translated for Sch-PAH patients, since this etiology was not included in the pivotal PAH trials. One of the most promising therapies for the treatment of PAH to emerge in recent years is selexipag, an oral IP receptor agonist, which acts on the prostacyclin pathway. The present study aims to evaluate the efficacy, safety and tolerability of selexipague for the treatment of schistosomiasis-associated pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic Sch-PAH. Sch-PAH diagnosis necessarily include the three criteria below

  1. Invasive confirmation of PAH, according to the criteria defined in the Pulmonary Hypertension Sixth World Symposium: mean pulmonary artery pressure higher than 20 mmHg, at rest, and the presence of pulmonary vascular resistance (PVR) equal to or greater than 3 W, and a pulmonary capillary pressure considered normal (equal to or lower than 15 mmHg (1)).
  2. At least one epidemiological criteria for chronic schistosomiasis: patient from a highly prevalent region for schistosomiasis or previous history of parasitic treatment for schistosomiasis or the presence of Schistosoma mansoni eggs in the patient's feces
  3. Evidence of long-term hepatosplenic involvement by schistosomiasis, via compatible ultrasound findings (peri-portal fibrosis or enlarged left lobe) All patients will necessarily already be receiving at least one specific treatment for PAH, either with phosphodiesterase V inhibitor or with an endothelin receptor antagonist, with a stable dose for at least 12 weeks before inclusion in the study.

     Exclusion Criteria:
* Patient without clinical condition to perform the 6-minute walk test
* Patient with gastro-intestinal bleeding for over 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance | 16 weeks

SECONDARY OUTCOMES:
FC | 16 weeks
  New York Heart Association Functional Class
6MWT | 16 weeks
  Lenght in the six minute walking distance test
BNP | 16 weeks
  Brain Natriuretic Peptide
HSP 70 | 16 weeks
  Heat shock protein 70

OTHER OUTCOMES:
ESC/ERS risk stratification category | 16 weeks
  ESC/ERS risk stratification category

CONTACTS AND LOCATIONS:
Overall Officials: Caio J Fernandes, PHD, Principal Investigator — USP
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No